CLINICAL TRIAL: NCT02378038
Title: A Phase II Study of PNT2258 in Patients With Richter's Transformation (RT)
Brief Title: PNT2258 for Treatment of Patients With Richter's Transformation (Brighton)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNT2258-04-Richter's
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Richter's Transformation
Keywords: PNT2258; Richter's Transformation; NHL; Non-Hodgkin's Lymphoma; Lymphoma; DLBCL; Diffuse Large B-cell Lymphoma; Lymphoma, Large B-cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, B-cell
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell | interventions — PNT100

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PNT2258 (Experimental): PNT2258 will be administered at 120 mg/m2 on days 1-5 of a 21-day cycle for 8 induction cycles followed by continuation phase therapy at a dose of 100 mg/m2 on days 1-4 of a 28-day cycle.
  Interventions: Drug: PNT2258

INTERVENTIONS:
Drug: PNT2258

SUMMARY:
This study is sponsored by Sierra Oncology, Inc. formerly ProNAi Therapeutics, Inc. It is a multi-center, single-arm, 2-stage, open-label phase II investigation of PNT2258 to characterize anti-tumor activity and collect safety data on patients with Richter's Transformation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Richter's transformation (RT) from chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL).
2. Availability of fresh or archived tumor tissue.
3. FDG PET-CT (disease) positive baseline scan with measurable disease.
4. ECOG performance status of 0-1.
5. Evidence of disease progression at study entry.
6. Discontinuation of prior anticancer therapy for ≥ 7 days prior to C1D1 and recovered to ≤ CTCAE grade 2 (or baseline) from any acute or chronic toxicity associated with prior therapy.
7. Must have previously received at least one prior chemotherapeutic regimen for RT.

   - Previously untreated RT patients deemed ineligible for, or that refuse, intensive chemotherapy are eligible.
8. Adequate bone marrow, renal, and hepatic function.
9. Normal Coagulation profile.
10. Agreement to use acceptable methods of contraception during the study and for ≥ 120 days after the last dose of PNT2258 if sexually active and able to bear or beget children.
11. Ability to participate in the clinical study for a minimum of at least 2 cycles (6 weeks).

Exclusion Criteria:

1. Concurrent non-hematologic malignancies requiring treatment.
2. No more than 2 prior regimens for DLBCL.
3. Hodgkin's variant of Richter's lymphoma, accelerated CLL, composite lymphoma, interdigitating dendritic cell sarcoma, sarcoma, EBV-associated lymphoma or prolymphocytic transformation.
4. Ongoing risk of bleeding.
5. CNS or leptomeningeal involvement of lymphoma
6. Concurrent clinically significant illness, medical condition, surgical history, physical finding, electrocardiogram or laboratory finding that, in the opinion of the investigator, could adversely affect the safety of the subject or impair the assessment of the study results.
7. Pregnancy or breast-feeding.
8. Previous exposure to PNT2258.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Klencke, MD, Study Chair — Sierra Oncology LLC - a GSK company
Locations (9):
- United States (9):
  - UC Irvine Medical Center, Orange, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Tyler Hematology Oncology, Tyler, Texas
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initiated in August 2015 and the first subject was enrolled on 27 October 2015. Enrollment was closed as of 07 June 2016. Subjects were enrolled at oncology clinics in the USA.
Groups:
- PNT2258: PNT2258 administered at 120 mg/m2 on days 1-5 of a 21-day cycle for 8 induction cycles followed by continuation phase therapy at a dose of 100 mg/m2 on days 1-4 of a 28-day cycle.
Period: Overall Study
Arm/Group | PNT2258
Started | 5
Completed | 0
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | PNT2258
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 73 [65 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Proportion of subjects with complete response (CR/CMR) or partial response (PR/PMR)
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | PNT2258
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Disease Control Rate
Description: Proportion of subjects with stable disease or better (CR/CMR, PR/PMR or SD/NMR)
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | PNT2258
Number analyzed (Participants) | 5
Participants | 0

3. Secondary Outcome: Duration of Overall Response
Time Frame: 2 months
Population: Analysis not performed as there were no responders.
Arm/Group | PNT2258
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Response
Time Frame: 2 months
Population: Analysis not performed as there were no responders.
Arm/Group | PNT2258
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression Free Survival
Time Frame: 2 months
Population: Analysis not performed as the study was terminated.
Arm/Group | PNT2258
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival
Time Frame: 2 months
Population: Analysis not performed as the study was terminated.
Arm/Group | PNT2258
Number analyzed (Participants) | 0

7. Secondary Outcome: Safety - Assessment of Adverse Events
Time Frame: 2 months
Measure: Number; unit: participants reporting at least 1 AE
Arm/Group | PNT2258
Number analyzed (Participants) | 5
participants reporting at least 1 AE | 5

ADVERSE EVENTS:
Time Frame: From the first dose of PNT2258 until 30 days after the last dose of PNT2258
Arm/Group | PNT2258
All-Cause Mortality (participants affected / at risk) | 2/5
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PNT2258 (N=5)
Atrial fibrillation (Cardiac disorders) | 1
Pyrexia (General disorders) | 1
Listeriosis (Infections and infestations) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 1
Disease progression (General disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PNT2258 (N=5)
Anaemia (Blood and lymphatic system disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Faecal incontinence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 2
Chills (General disorders) | 1
Early satiety (General disorders) | 1
Fatigue (General disorders) | 3
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 1
Cytomegalovirus viraemia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Embolism (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination of enrollment, and thus very few subjects were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days